CLINICAL TRIAL: NCT06124313
Title: A Single Group Study to Evaluate the Effects of a Vaginal Probiotic on Vaginal and Digestive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rael (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20337
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome; Vaginal Health
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will take one capsule of the test product every day, with water.
  Interventions: Dietary Supplement: Vaginal Probiotic

INTERVENTIONS:
Dietary Supplement: Vaginal Probiotic — This product contains:
  Probiotic Blend - 5 Strains Lactobacillus acidophilus Lactobacillus rhamnosus Lactobacillus gasseri Lactobacillus acidophilus (NCFM) Lactobacillus casei

SUMMARY:
This is a virtual single-group study that will last 12 weeks. Participants will take 1 capsule every day, with water. Questionnaires will be completed at baseline, 2 weeks, 4 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40
2. Self-reported concerns with vaginal odor, itchiness, dryness, or discharge
3. Self-reported issues associated with bacterial Vaginosis, reporting three of the following symptoms:

   * Unusual vaginal discharge ( thin, grayish-white or milky discharge that has a strong, fishy odor)
   * Changes in vaginal odor (i.e. An unpleasant "fishy" odor)
   * Vaginal itching or irritation
   * Discomfort or burning sensation during urination
4. Self-reported symptoms associated with irritable bowel syndrome (IBS), including three of the following symptoms:

   * Abdominal pain or discomfort
   * Changes in bowel habits i.e. diarrhea, constipation, or a combination of both.
   * Bloating
   * Gas or flatulence
   * Changes in stool appearance
   * Mucus in the stool
5. Generally healthy - don't live with any uncontrolled chronic diseases
6. Willing to avoid the use of any intra-vaginal products (such as vaginal creams, gels, or medications) as well as suppositories during the study product use

Exclusion Criteria:

1. Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
2. Planning to undergo any procedure related to their reproductive health.
3. Started any new medications or supplements that target vaginal health or IBS in the past 3 months.
4. Anyone with known severe allergic reactions
5. Women who are pregnant, breastfeeding, or attempting to become pregnant
6. Unwilling to follow the study protocol
7. Anyone with a history of vaginal, cervical, vulvar, uterine, or ovarian cancer
8. Anyone who has changed or stopped taking hormonal birth control in the last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms of bacterial vaginosis. | Baseline to Week 12
  Participants will complete self-reported questionnaires reporting on incidence and severity of symptoms of bacterial vaginosis.
Changes in vaginal odor. | Baseline to Week 12
  Participants will complete self-reported questionnaires reporting their perceptions of their vaginal odor. Responses will be gathered on a 5-point Likert scale, with 0= the most favorable severe and 5= the least favorable response.
Changes in vaginal itchiness. | Baseline to Week 12
  Participants will complete self-reported questionnaires reporting the severity of vaginal itching. Responses will be gathered on a 5-point Likert scale, with 0= the least severe and 5= most severe response.
Changes in vaginal discharge. | Baseline to Week 12
  Participants will complete self-reported questionnaires reporting their perceptions of their vaginal discharge. Responses will be gathered on a 5-point Likert scale, with 0= the most favorable severe and 5= the least favorable response.
Changes in vaginal dryness. | Baseline to Week 12
  Participants will complete self-reported questionnaires reporting the severity of vaginal dryness. Responses will be gathered on a 5-point Likert scale, with 0= the least severe and 5= most severe response.

SECONDARY OUTCOMES:
Changes in scores on the Gastrointestinal Symptom Rating Scale (GSRS). | Baseline to Week 12
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Changes in scores on the Bristol Stool Chart. | Baseline to Week 12
  On the Bristol Stool Chart, stools are assigned a number from 1 to 7, from hardest to loosest. Normal stools are those in the middle of the chart, in the 3 to 4 range

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided